CLINICAL TRIAL: NCT06766071
Title: The Texas A&M Interprofessional Pharmacogenomics PILOT Whole Genome Sequencing (WGS) Cohort
Brief Title: IPGx PILOT Whole Genome Sequencing Extension Cohort
Status: Recruiting | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY2024-0724
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-09

CONDITIONS: Adverse Drug Reaction (ADR); Polypharmacy Patients
Keywords: whole genome sequencing
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Biospecimen Retention: Samples With DNA — Blood, urine, and cheek swab sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator's primary aim is to evaluate polypharmacy-associated adverse drug reactions (ADR) in a pilot study of at-risk patients using state-of-the-art pharmacogenomic technology and to use this information to make recommendations for optimization of pharmacotherapy regimens. The data from the pilot cohort will be used to optimize and integrate a customized electronic decision support (clinical semantic network; CSN) dashboard to identify drug regimens that should be modified, replaced, or discontinued. A secondary objective of the pilot study is to evaluate the capacity/saturation of CYP P450 enzymatic pathways in polypharmacy patients. A third objective is to determine the feasibility of the planned informatics workflows between the CLIA lab, the EMR, and the Family Medicine Practice including Whole Genome Sequencing (WGS).

DETAILED DESCRIPTION:
The investigators are concerned with patient safety and ADRs as these areas of clinical practice represent significant causes of death, ahead of many of the better recognized acute and chronic causes of mortality. While prescribing medicines can have life-altering benefits, a more precise way of choosing among the options on a formulary continues to lag behind existing technologies. A person's drug response can vary by means of drug-drug or drug-food interactions, as well as by sex, age, and disease status. Large interpersonal variabilities of up to 1000-fold exist in response to the same dose of a given medication. Genetic polymorphisms help define pharmacokinetic and pharmacodynamic profiles, but these insights have not yet been consistently incorporated into clinical practice and standards of care. Several medication management programs have appeared in recent years, but these are mainly geared toward adherence, with only limited incorporation of pharmacogenomics-based medication management. Precision medicine advocates that one size does not fit all medical care. How might the provision of care get closer to the bullseye in polychronic disease management, and the management of polypharmacy?

There exists a polypharmacy crisis in the United States that is large in scope, especially among the older populations who often have diminishing renal and hepatic functions. The prevalence of potential hepatic cytochrome enzyme-mediated drug-drug interactions was estimated to be as high as 80% in one study with elder adults considered to be more susceptible to problematic drug interactions. Conventionally, polypharmacy refers to taking five or more medications concurrently. An estimated 15 million patients 65 or older have been identified as facing the challenge. Polypharmacy patients often have at least two comorbid chronic diseases, and nearly 50% of older adults are using at least one medication that is not necessary. Hospitalized patients average five to eight medications, and the number surpasses nine in 40% of nursing home residents. In a study of patients with cognitive decline or mild Alzheimer's disease, 88% of these patients met polypharmacy criteria, with anticholinergic cognitive burden, drug-drug interactions, and drug-gene interactions all prevalent issues in these populations. In an increasing number of extreme cases, polypharmacy can approximate 20 drugs posing risks for adverse drug outcomes that equal nearly 100%. The greater the number of medications in a regimen, the higher the risk to patient safety and compromised clinical outcomes. One in twenty polypharmacy outpatients seek medical care for ADRs. Polypharmacy has also been associated with hospitalizations among the elderly. Polypharmacy is associated with decreased medication adherence, nutrition, urinary incontinence, reduced activities of daily living, and loss of physical and cognitive functions. Increased falls occur along with accompanying morbidity and mortality. Financially, the impact of polypharmacy has been associated with a 30% increase in health care expenditures, and a major factor in ultrahigh healthcare utilizers. Analysis of the Observational Health Data Sciences and Informatics data set showed that 10% of diabetes patients, 24% of hypertension patients, and 11% of depression patients followed a treatment pathway that was unique among a population of 250 million cases, illustrating the need for electronic decision support to flag drug interactions resulting from patient specific care plans and implement corrective measures.

Electronic health records continue to fall short regarding their level of interoperability, with significant deficiencies enabling a care plan and medication management that can draw data and decision support from across the provider continuum. This is a suboptimal situation in the provision and refinement of precision and personalized medical care. The clinical burden of polypharmacy and medication reconciliation often impacts primary care clinicians who may not have the necessary data at the point of service, a nidus for polypharmacy management problems. Innovative approaches to managing the polypharmacy challenge include the creation of medical management clinics with focused efforts on mitigating the cost and healthcare burden of polypharmacy and to systematically evaluate the incremental clinical changes that accompany medication alterations, modification or discontinuation where indicated.

Utilizing an interprofessional care team that includes physicians, pharmacists, nurses, case coordinators, along with telemedicine and digital tools, the investigators can engage patients and garner information such as phenotypic, functional, and social determinants of disease profiles. These data can be entered as computable actionable data prior to a visit in order to better track what happens in- between visits (adherence to the care plan, or lack thereof). The investigators posit that this information is as important as what happens at an appointment, and this is especially true in clinical cases of polypharmacy. In the end, this information can become more readily available to both patient and provider utilizing the Interprofessional Pharmacogenomics (IPGx) care model.

The investigators are developing a care decision support protocol and pharmacogenomic/ pharmacokinetic dashboards that augment the capacity for primary care clinicians to manage medication more precisely for individual cases and that is minimally disruptive. Additionally, interoperability between electronic medical records, clinical decision support (CDS) and genomic test data formats remains a barrier for reuse of PGx tests and implementation of whole genome and whole exome sequencing across time and different healthcare providers. These efforts will inform the feasibility of using whole genome sequencing (research use only under this study protocol) across the informatics platforms used in the IPGx care model.

The dashboards will be useful to providers and patients, helping to identify clinical cases where there might be benefit from proactive medication management to identify those who may not respond and those at heightened risk of ADRs. The dashboards would be informed by a growing library of clinical cases with a clinical data warehouse. The dashboard would generate and iteratively refine novel care decision trees (algorithms) centered on medication management. The data structure and care protocol are designed to enable concomitant and longitudinal observation (research) of the clinical activities toward validation of the ActX CDS and dashboards as a useful tool for patient-centric clinical research. The ideal databank will include drug blood levels (not relevant to this PILOT), drug list and other relevant modifier data that may impact medication use and effectiveness. This approach would also provide a means to learn more about drug adherence and help to systematically identify patients who may be candidates for a pharmacogenomic evaluation and longer-term participation in a medication management program.

Specific questions that this GENERALIZED approach might inform:

Does a drug level near zero mean non-adherence, or is the patient metabolizing a drug extensively such that blood or urine levels become undetectable after administration? The phenotypic questionnaire coupled with drug blood or urine level measurements will answer that question.

Is a protocol needed to determine when to order a pharmacogenomic test? The investigator's data platform, powered by the ActX platform, can validate the clinical and cost-effectiveness of those decisions.

What is the best use pharmacogenomic data? If a patient has had a pharmacogenomic test, blood or urine drug levels might help refine knowledge about the metabolic activity for pertinent enzymatic pathways and help craft key questions to identify what constitutes an overloaded CYP P450 pathway in the setting of polypharmacy.

ADRs might be preventable in the psychotropic domain by applying the knowledge derived from a medication management consultation. For instance, in the case of antidepressants, weeks may go by before a clinical response can be evaluated after initiating medication based on standard dosing and trial and error. In a precision medication management scenario, the provider would know at the outset if the patient were an ultra-rapid metabolizer for a relevant CYP P450 enzymatic pathway and be better equipped to identify the drug of choice and to optimize dose titration. If the clinical dashboard reveals a patient that is receiving several medications competing for a common pathway, proper medication adjustments can also be made, as needed.

The ActX to be used here is a clinical decision support system containing millions of interrelated variant-drug concepts that arc with each other to create a knowledge network. As data is entered, weighted arcs are used to build clinical decision support and differential diagnoses. This provides a potentially strong environment for a pharmacogenomic profile to create a precision drug and dosing regimen tool while taking advantage of clinical workflows currently in practice. The pharmacogenomic dashboard is contained within the ActX platform.

Compare and contrast WGS and Genotyping

The ActX test is a genotyping test conducted in a CAP/CLIA-compliant laboratory for complex lab-developed tests (LDTs) to ensure that results can be used for clinical decision-making within the LDT regulatory framework. This type of test examines a limited number of features in the human genome, specifically just under 400 known genetic variants with clinical significance. The results from the ActX test will be returned to the provider and discussed with patients. Whole Genome Sequencing (WGS) provides a complete comprehensive inventory of the entire human genome, which consists of approximately 4 billion base pairs. While WGS can be performed under CAP/CLIA regulations for clinical decision-making, the testing laboratory we will be using will conduct a Research Use Only (RUO) test and WILL NOT be an LDT. As a result, WGS results will not be provided to healthcare providers or patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals taking 5 or more medications, including over the counter drugs, supplements, natural products, cannabis produces, or other recreational drugs.
* Ability to give and comprehend the consent process.
* Consent to donate urine samples, genetic data through buccal swabs and blood samples, and undergo a comprehensive history and physical examination.
* All genders
* Age 18-100

Exclusion Criteria:

* Subject has been diagnosed or is being treated for any cancer other than basal cell cancer in the last 5 years. Patients with metastatic melanoma in the last 5 years will be excluded.
* Admitted to hospice.
* Patient has ever been diagnosed with Hepatitis B or C.
* Patient has ever been diagnosed with active liver disease, hepatomegaly, grossly abnormal liver function. Meld score >10, ALT, or AST >100U/L or an AST/ALT ratio >2
* Patients taking imidazole antifungal medication.
* Declines to participate or interact with staff/share their medical status.
* A diagnosis of Alzheimer's disease or related dementias in a medical record indicates a progressive, debilitating condition that impairs memory, thought processes, and functioning.
* Pregnant patients will be excluded.
* Individuals who are unable or unwilling to provide consent will be excluded.
* Unable to verbally communicate and comprehend English language.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to recruit at most 50 volunteers from the Texas A&M affiliated community health family medicine program.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacogenomic genotype with corresponding ADR phenotype | 180 days
  Patients will be referred to the Texas A&M Interprofessional Pharmacogenomics Clinic (IPGx) by their primary care physicians to evaluate genotyping and ADR. Clinical staff will obtain a buccal swab to collect DNA for a pharmacogenomic evaluation pursuant to the sample collection kits from the CLIA lab, which will occur at the start of the study period. Blood chemistry will be taken from the EMR.

SECONDARY OUTCOMES:
Emergency department visits | 180 days
  A secondary objective of the pilot study is to evaluate & monitor the frequency of Emergency department visits.

OTHER OUTCOMES:
Drug-drug interactions, drug gene interactions, drug-drug-gene interactions | 180 days
  An assessment at the IPGx will start with the pharmacist or physician doing a pharmacologic consultation to evaluate medications or other drugs currently being used by the patient and to identify any potential issues related to toxicity, drug interactions, or side effects that might be relevant to the clinical presentation.
Frequency and nature of ADRs on the Naranjo Scale | 180 days
  Patients will be referred to the Texas A&M Interprofessional Pharmacogenomics Clinic (IPGx) by their primary care physicians. A physician or ambulatory pharmacist in the IPGx clinic or Family Care Clinic will obtain a complete medical history, physical examination, and validate the patient's current concomitant medication list at the IPGx during the office visit. Patient medical information would be input into the ActX platform, which functions as a computable EHR medical record analysis, evaluation of polypharmacy status, and monitoring of ADRs using the Naranjo Scale (19) will be conducted for the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M Family Care, Bryan, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT06766071/Prot_000.pdf